CLINICAL TRIAL: NCT02917746
Title: TOPical Imiquimod Treatment of High-grade Cervical Intraepithelial Neoplasia, a Multicenter, Open-label, Non-randomized, Controlled Study (TOPIC-3 Study)
Brief Title: Imiquimod Treatment of High-grade CIN
Acronym: TOPIC-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Clinical Trial Center Maastricht B.V. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL 57849.068.16
Record Dates: First submitted 2016-09-16; First posted 2016-09-28 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-05

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical intraepithelial neoplasia; Imiquimod; Treatment; Predictive biomarkers
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imiquimod treatment arm (Experimental): Treatment by vaginal imiquimod cream during 16 weeks.
  Interventions: Drug: Imiquimod
- Standard treatment arm (Active Comparator): Treatment by large loop excision of the transformation zone.
  Interventions: Procedure: Large Loop Excision of the Transformation Zone

INTERVENTIONS:
Drug: Imiquimod — Patients in this group are treated with vaginal imiquimod cream during 16 weeks. A control colposcopy with diagnostic biopsies will be performed after 10 weeks to rule out disease progression. A final colposcopy with diagnostic biopsies will be performed after 20 weeks to evaluate disease efficacy.
  Arms: Imiquimod treatment arm
Procedure: Large Loop Excision of the Transformation Zone — Patients in this group are treated with LLETZ.
  Arms: Standard treatment arm

SUMMARY:
This multi-center, open-label, non-randomized controlled intervention study aims to investigate the treatment efficacy, side-effects and quality of life associated with imiquimod treatment of high-grade CIN lesions, as an alternative to surgical treatment by Large Loop Excision of the Transformation Zone (LLETZ). Non-surgical treatment may prevent side-effects associated with surgical treatment, such as premature birth in subsequent pregnancies. The study hypothesis is that approximately 75% of patients with high-grade CIN will be adequately treated with imiquimod.

120 women with a histological diagnosis of CIN2 or CIN3 will be included and allocated to one of two treatment arms according to their preference:

1. Imiquimod treatment arm(60 patients). Patients in this group are treated with vaginal imiquimod 5% cream during 16 weeks.
2. Standard treatment arm (60 patients). Patients in this group will undergo LLETZ treatment.

DETAILED DESCRIPTION:
Cervical Intraepithelial Neoplasia (CIN) is the premalignant condition of cervical cancer. The standard treatment of histologically confirmed CIN2-3 is surgical excision by large loop excision of the transformation zone (LLETZ). This procedure has potential complications, such as hemorrhage, infection and preterm birth in subsequent pregnancies. For this reason, non-invasive therapies are needed. Imiquimod cream has been studied as a non-invasive treatment alternative in high-grade CIN, but evidence on treatment efficacy is limited and evidence on disease recurrence and quality of life during and after treatment is lacking. One RCT has been performed and shows that treatment of high-grade CIN with vaginal imiquimod cream leads to disease regression in 73%. Side-effects were generally mild, but common. A recent survey among gynecologists and a patient preference study indicate that imiquimod treatment of high-grade CIN is mainly preferred by a selected population of women with a future pregnancy wish. These women accept a lower treatment efficacy and higher rates of side-effects from imiquimod treatment in order to prevent future preterm birth caused by LLETZ treatment. Ideally, those women with a high probability of successful treatment would be selected.

The objective of this study is to investigate the treatment efficacy, side-effects and quality of life associated with imiquimod treatment of high-grade CIN lesions in a selected population of patients who prefer imiquimod treatment instead of LLETZ. The study also aims to identify predictive biomarkers clinical response to imiquimod treatment, in order to select patients in which good treatment response is expected.

The study design is a multicenter, open-label, non-randomized controlled intervention study. 120 women with a histological diagnosis of CIN2 or CIN3 will be included and allocated to one of two treatment arms according to their preference:

1. Imiquimod treatment arm(60 patients). Patients in this group are treated with vaginal imiquimod 5% cream during 16 weeks.
2. Standard treatment arm (60 patients). Patients in this group will undergo LLETZ treatment.

A control colposcopy will be performed after 10 weeks for the imiquimod group. In case of progressive disease, the treatment will be ended and LLETZ will be performed as treatment. For patients in which the treatment is continued, treatment efficacy will be evaluated after 20 weeks, by colposcopy with diagnostic biopsies. Statistical analysis will be performed based on an intention-to-treat analysis.

The primary study endpoints are:

* Treatment efficacy of imiquimod and LLETZ treatment, defined as regression to CIN1 or less after 20 weeks for imiquimod and no need for additional therapy within 6 months for LLETZ treatment.
* Identification of predictive biomarkers for the efficacy of imiquimod treatment in the individual patient, based on biomarkers reflecting host, virus and cellular factors.

Secondary study endpoints are:

* Side effects of imiquimod therapy and LLETZ therapy.
* Disease recurrence at 6, 12 and 24 months follow-up.
* Quality of life (QoL) before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* de novo CIN2 or CIN3 lesion, histologically confirmed by diagnostic biopsy
* age of 18 years or older

Exclusion Criteria:

* previous histologically confirmed high-grade CIN (CIN 2-3)
* concomitant vulvar and/or vaginal intraepithelial neoplasia
* previous cervical malignancy
* current malignant disease
* immunodeficiency (including HIV/AIDS and immunodepressive medication)
* pregnancy or lactation
* legal incapability

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy of imiquimod 5% cream for the treatment of CIN2-3 lesions, compared to LLETZ treatment, in selected populations. | 6 months
  Treatment efficacy for the imiquimod group is defined as regression to CIN 1 or less at 20 weeks follow-up. Treatment efficacy for the standard treatment group is defined as no need for additional treatment within 6 months after LLETZ treatment.
Identification of predictive biomarkers for treatment efficacy of imiquimod in the individual patient. | Baseline (T=0)
  Histological biomarkers will be identified in the cervical biopsies performed at baseline.

SECONDARY OUTCOMES:
Side effects of imiquimod therapy and LLETZ therapy. | 20 weeks
  Scored by the Common Terminology Criteria for Adverse Events guidelines.
Disease recurrence | 6, 12 and 24 months
  Defined as abnormal cervical cytology for all treatment groups.
General health-related Quality of life (QoL) before, during and after treatment | Baseline, 20 weeks and 1 year
  Medical Outcomes Study 36-Item Short-Form General Health Survey (RAND 36)
Cancer specific Quality of Life, during and after treatment | Baseline, 20 weeks and 1 year
  European Organization for Research and Treatment of Cancer (EORTC) quality-of-life questionnaire: QLQ-C30
Cervical cancer specific Quality of life (QoL), during and after treatment | Baseline, 20 weeks and 1 year
  European Organization for Research and Treatment of Cancer (EORTC) quality-of-life questionnaire: QLQ-CX24

CONTACTS AND LOCATIONS:
Overall Officials: A.J. Kruse, MD, PhD, Study Director — Maastricht University Medical Center
Locations (3):
- Netherlands (3):
  - Meander Medical Center, Amersfoort
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crane JM. Pregnancy outcome after loop electrosurgical excision procedure: a systematic review. Obstet Gynecol. 2003 Nov;102(5 Pt 1):1058-62. doi: 10.1016/s0029-7844(03)00741-5. PMID 14672487
- [Background] Kyrgiou M, Koliopoulos G, Martin-Hirsch P, Arbyn M, Prendiville W, Paraskevaidis E. Obstetric outcomes after conservative treatment for intraepithelial or early invasive cervical lesions: systematic review and meta-analysis. Lancet. 2006 Feb 11;367(9509):489-98. doi: 10.1016/S0140-6736(06)68181-6. PMID 16473126
- [Background] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404
- [Background] Pachman DR, Barton DL, Clayton AC, McGovern RM, Jefferies JA, Novotny PJ, Sloan JA, Loprinzi CL, Gostout BS. Randomized clinical trial of imiquimod: an adjunct to treating cervical dysplasia. Am J Obstet Gynecol. 2012 Jan;206(1):42.e1-7. doi: 10.1016/j.ajog.2011.06.105. Epub 2011 Jul 13. PMID 21907959
- [Background] Lin CT, Qiu JT, Wang CJ, Chang SD, Tang YH, Wu PJ, Jung SM, Huang CC, Chou HH, Jao MS, Lai CH. Topical imiquimod treatment for human papillomavirus infection in patients with and without cervical/vaginal intraepithelial neoplasia. Taiwan J Obstet Gynecol. 2012 Dec;51(4):533-8. doi: 10.1016/j.tjog.2012.09.006. PMID 23276555
- [Background] Koeneman MM, van de Sande AJ, van Beekhuizen HJ, Gerestein KG, van de Laar R, Kruitwagen RF, Kruse AJ. Physicians' Awareness, Attitudes, and Experiences Regarding Imiquimod Treatment of Vaginal and Cervical Intraepithelial Neoplasia. J Low Genit Tract Dis. 2016 Jan;20(1):75-9. doi: 10.1097/LGT.0000000000000158. PMID 26579838
- [Derived] Koeneman MM, Kruse AJ, Kooreman LF, Zur Hausen A, Hopman AH, Sep SJ, Van Gorp T, Slangen BF, van Beekhuizen HJ, van de Sande AJ, Gerestein CG, Nijman HW, Kruitwagen RF. Preliminary stop of the TOPical Imiquimod treatment of high-grade Cervical intraepithelial neoplasia (TOPIC) trial. BMC Cancer. 2017 Feb 7;17(1):110. doi: 10.1186/s12885-017-3108-9. PMID 28173776